CLINICAL TRIAL: NCT02754570
Title: The Diurnal and Nocturnal Effect of Pilocarpine on Intraocular Pressure and Ocular Perfusion Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-1972; UL1TR001082 (NIH)
Record Dates: First submitted 2016-04-20; First posted 2016-04-28 (Estimated); Results first posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-10

CONDITIONS: Glaucoma, Open-angle; Hypertension, Ocular
Keywords: Open-angle glaucoma; Ocular hypertension; Latanoprost; Pilocarpine
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Pilocarpine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pilocarpine group (Experimental): Subjects with open-angle glaucoma and ocular hypertension that are currently taking latanoprost
  Interventions: Drug: Pilocarpine

INTERVENTIONS:
Drug: Pilocarpine — Pilocarpine will be administered 4 times in addition to latanoprost.
  Other Names: Pilocarpine Hydrochloride

SUMMARY:
The aim of this study will be to determine the effects of pilocarpine as an adjunct medication to latanoprost monotherapy at multiple intervals throughout a 24-hour period and compare these effects to latanoprost alone.

DETAILED DESCRIPTION:
This study plans to learn more about the effect of pilocarpine on intraocular pressure and ocular perfusion pressure for a full twenty-four hour period.

In this study, the investigators seek to better characterize the knowledge base of the intraocular pressure (IOP) lowering effects of pilocarpine in patients with open angle glaucoma or ocular hypertension who are currently taking latanoprost. The goal is to define the potential additive effect of pilocarpine throughout a 24-hour period, not only for IOP, but for ocular perfusion pressure (defined as 2/3[diastolicBP + 1/3(systolicBP - diastolicBP)] - IOP). These data will allow to expand current knowledge of the effects of pilocarpine and help determine if this medication has a useful role as an adjunctive treatment in glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Current confirmed diagnosis of:

  * open angle glaucoma, or
  * ocular hypertension including pigment dispersion glaucoma, and
  * pseudoexfoliation glaucoma.
* Current use of topical latanoprost once a day in both eyes for at least 6 weeks
* any race/ethnicity

Exclusion Criteria:

* Females who are currently pregnant or planning to become pregnant during the study period
* Diagnosis of any other form of glaucoma other than open-angle
* Intraocular pressure readings of <14mmHg in either eye when measured during routine office visit in the past 12 months.
* Schaffer angle grade < 2 in either eye by gonioscopy
* Intraocular surgery within 6 months or laser within 3 months
* History of retinal tear or detachment in either eye
* Active iritis in either eye as determined by most recent eye examination
* Patients who smoke or have irregular daily sleep patterns
* Patients who have started or changed glucocorticoids therapy in the last 3 months
* Patients who are currently using medical or recreational marijuana
* Any use of a non-FDA approved medication for glaucoma in the last 3 months

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-07; Primary Completion 2017-12 (Actual); Study Completion 2018-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Seibold, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver Eye Hospital, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pilocarpine Group: Subjects with open-angle glaucoma and ocular hypertension.
  Pilocarpine: Pilocarpine will be administered 4 times in addition to latanoprost.
Period: Overall Study
Arm/Group | Pilocarpine Group
Started | 27
Visits 1 and 2 (PGA Only) | 27
Visit 3 (PGA + Pilocarpine) | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pilocarpine Group
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 19
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 27
Diagnosis [Count of Participants; unit: Participants]
  Primary Open Angle Glaucoma | 21
  Ocular Hypertension | 4
  Pseudoexfoliation Glaucoma | 2
Lens Status [Count of Participants; unit: Participants]
  Phakic | 19
  Pseudophakic | 8
Prior Laser Surgery [Count of Participants; unit: Participants]
  Laser Peripheral Iridotomy | 5
  Selective Laser Trabeculoplasty | 3
  No Prior Laser | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure From Baseline at Visit 3
Description: Subjects will be enrolled at the first visit. Patients already on latanoprost may proceed immediately with the second visit. Patients on a different prostaglandin analog medication will be switched to latanoprost for at least 6 weeks. At second visit, intraocular pressure and blood pressure will be measured every 2 hours for a 24-hour period. At any point over the next 4 weeks, another 24-hour visit will be performed. This time, a dose of pilocarpine 2% will be administered at 4 different times in addition to the latanoprost . As before, intraocular pressure and blood pressure will be measured every 2 hours. After visit 3, subjects will return to their prior treatment regimen. Change in the intraocular pressure from the second and the third visit will be determined. 8 diurnal readings and 4 nocturnal readings were averaged separately during both Visit 2 for the PGA Monotherapy and Visit 3 for Pilocarpine+PGA
Time Frame: Two 24-hour visits: Baseline/Visit 2; Up to week 4/Visit 3
Population: Patients who are using a prostaglandin analog (PGA) will be monitored at visit two. At visit 3, pilocarpine will be added four times per day to the PGA therapy.
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Pilocarpine Group: Subjects with open-angle glaucoma, ocular hypertension or pseudoexfoliation glaucoma.
  Pilocarpine: Pilocarpine will be administered 4 times in addition to latanoprost or brimonidine
Arm/Group | Pilocarpine Group
Number analyzed (Participants) | 27
mmHg
  Visit 2: Nocturnal PGA | 21.1 (0.7)
  Visit 2: Diurnal PGA | 18.2 (0.5)
  Visit 3: Nocturnal PGA | 20.0 (0.6)
  Visit 3: Diurnal PGA | 17.1 (0.4)

2. Secondary Outcome: Change in Ocular Perfusion Pressure
Description: Ocular perfusion pressure will calculated from the intraocular pressure and blood pressure measurements. At Baseline/Visit 2, intraocular pressure and blood pressure will be measured every 2 hours for a 24-hour period. At any point over the next 4 weeks, another 24-hour visit (Visit 3) will be performed. This time, a dose of pilocarpine 2% will be administered at 4 different times in addition to the latanoprost (PGA monotherapy). As before, intraocular pressure and blood pressure will be measured every 2 hours. 8 diurnal readings and 4 nocturnal readings were averaged separately during both Visit 2 for the PGA Monotherapy and Visit 3 for Pilocarpine+PGA
Time Frame: Two 24-hour visits: Baseline/Visit 2; Up to week 4/Visit 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Pilocarpine Group: Subjects with open-angle glaucoma, ocular hypertension or psuedoexfoliation glaucoma.
  Pilocarpine: Pilocarpine will be administered 4 times in addition to latanoprost.
Arm/Group | Pilocarpine Group
Number analyzed (Participants) | 27
mmHg
  Visit 2: Diurnal Ocular Perfusion Pressure | 44.12 (1.2)
  Visit 2: Nocturnal Ocular Perfusion Pressure | 37.2 (1.3)
  Visit 2: Diurnal Systolic Blood Pressure | 132.5 (2.8)
  Visit 2: Nocturnal Systolic Blood Pressure | 125.8 (2.9)
  Visit 3: Diurnal Ocular Perfusion Pressure | 44.3 (1.1)
  Visit 3: Nocturnal Ocular Profusion Pressure | 37.1 (1.2)
  Visit 3: Diurnal Systolic Blood Pressure | 130.8 (2.9)
  Visit 3: Nocturnal Systolic Blood Pressure | 122.7 (2.9)

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Pilocarpine Group: Subjects with open-angle glaucoma, ocular hypertension or pseudoexfoliation glaucoma.
  Pilocarpine: Pilocarpine will be administered 4 times in addition to latanoprost.
- PGA Monotherapy: Subjects with open-angle glaucoma, ocular hypertension or pseudoexfoliation glaucoma.
  PGA: Latanoprost or Bimatoprost administered one time per day.
Arm/Group | Pilocarpine Group | PGA Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT02754570/Prot_SAP_000.pdf